CLINICAL TRIAL: NCT06288477
Title: Clinical and Radiographic Evaluation of Vital Pulpotomy Techniques in Primary Molars Using of Premixed Bioactive Bioceramic MTA (Neo-putty) as a Novel Pulpotomy Medication Versus Formocresol: A Randomized Clinical Trial.
Brief Title: Clinical and Radiographic Evaluation of Vital Pulpotomy Techniques in Primary Molars Using of Premixed Bioactive Bioceramic MTA (Neo-putty) as a Novel Pulpotomy Medication Versus Formocresol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October University for Modern Sciences and Arts (Other)
Responsible Party: Principal Investigator, Marwa Ahmed Salmoon, Principal Investigator, October University for Modern Sciences and Arts
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-2
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Vital; Pulpotomy; Techniques

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- full-strength FC (Active Comparator): Formocresol pulpotomy is one of the most common procedure in cases of mechanical and carious exposure in primary teeth.
  Interventions: Drug: A cotton pellet moistened with full-strength FC
- Neo-Putty® (Experimental): Neo-Putty® as dressing agents in pulpotomized primary molars. NeoPUTTY® is composed of extremely fine inorganic tricalcium/dicalcium silicate powders in a water-free organic liquid and contains tantalum oxide as the radiopacifying agent.
  Interventions: Drug: Neo-Putty

INTERVENTIONS:
Drug: A cotton pellet moistened with full-strength FC — A cotton pellet moistened with full-strength FC will be placed for 5 minutes on the amputated pulp, after reaching hemostasis. The pulp stumps will be then covered by IRM (Intermediate Restorative Material).
  Arms: full-strength FC
Drug: Neo-Putty — Following removal of the coronal pulp with a round bur and hemostasis, the pulp stumps in the study group will be covered with Neo-Putty ® according to the manufacturer's instructions. Neo-Putty will be placed in the prepared cavity, and then covered with a reinforced Zinc Oxide-Eugenol (IRM, Bayer-Leverkussen, Germany).
  Arms: Neo-Putty®

SUMMARY:
Despite the benefit of formocresol, there are toxic effects allergic reactions and local soft and hard tissue necrosis have been reported when such formaldehyde compounds were used clinically, however, the adverse effect of the clinically used of this compound are not widely reported. It has been stated that it has a side effect on the permanent successor although it results as a successful technique for the treatment of the primary teeth

DETAILED DESCRIPTION:
The rationale for conducting the research:

Nowadays, the introduction of new Bio-inductive materials resulted in the shift of the concept of preservation of radicular pulp tissue to regeneration. Restoration of the anatomical continuity of damaged tissue and disturbed functional status of the radicular pulp tissue require an appropriate method of wound healing which includes well-organized, biochemical and cellular events, leading to the growth and regeneration of injured radicular tissue in a special manner.

A higher standard in bioactive bioceramic putty as manufacture claimed the Neo-Putty® NuSmile is a bioactive bioceramic premixed root and pulp treatment with superior handling properties, promoting hydroxyapatite formation to support the healing process. Neo-Putty® is a premixed bioactive bioceramic root & pulp treatment consisting of an extremely fine, inorganic powder of tricalcium/dicalcium silicate in a water free organic liquid. The product is packaged ready to use. No mixing is required. Neo-Putty® is designed to set in vivo in the presence of moisture from the surrounding tissues. Considering the limitations of these data, we are conduction this clinical trial. The outcomes of this study will have a substantial impact on clinical practice for pediatric patients, as well as patient care, around the world.

Aim of the study:

This randomized clinical trial study will assess clinically and radiographically, the effect of Neo-Putty® as a pulp medicament following coronal pulp amputation in children's primary molars with carious pulp exposure in comparison to Formocresol (FC).

Research question:

Is the pulpotomy procedure in primary molars using premixed Bioactive bioceramic MTA (Neo-putty) more clinically successful than Formocresol?

PICOS:

P: Carious primary molars with no spontaneous or provoked pain (vital primary molars) I: Neo-Putty® as dressing agents in pulpotomized primary molars C: Formocresol Pulpotomy (FC) O: Clinical Success S: In-Vivo Study II. Methods

Study Design:

Study Type: Interventional (Clinical Trial) Estimated Enrolment: 88 participants Allocation: Randomized Intervention Model: Parallel Assignment Primary Purpose: Treatment Official Title: Clinical and Radiographic Evaluation of Vital Pulpotomy in Primary Molars using of premixed Bioactive bioceramic MTA (Neo-putty) as a Novel Pulpotomy Medication versus Formocresol: A Randomized Clinical Trial. Estimated Study Start Date: December 2023 Estimated Primary Completion Date: January 2024

Trial design:

The study is a randomized clinical trial (RCT) where 2 arm parallel groups with a 1:1 allocation ratio were compared. The child participants and the legal guardian of each participating child and the statistician were blinded.

Interventions In the control group: a cotton pellet moistened with full-strength FC will be placed for 5 minutes on the amputated pulp, after reaching hemostasis. The pulp stumps will be then covered by IRM.

In the Intervention group:

Neo-Putty® as dressing agents in pulpotomized primary molars. Following removal of the coronal pulp with a round bur and hemostasis, the pulp stumps in the study group will be covered with Neo-Putty ® according to the manufacturer's instructions. Neo-Putty will be placed in the prepared cavity, and then covered with a reinforced Zinc Oxide-Eugenol (IRM, Bayer-Leverkussen, Germany).

Outcome Measures:

1. Primary outcome: Clinical success [Time Frame: 12 months].

* Success clinically and radiographically will assess by the number of participants with symptoms-free and no peri-radicular pathology (at 3,6,9and 12 months)
* No clinical or radiographic evidence of pulp degeneration, such as spontaneous pain, excessive bleeding from the root canal, internal root resorption, inter-radicular and/or periapical bone destruction, swelling, or sinus tract.

ELIGIBILITY:
Criteria The eligibility criteria were set according to the guidelines of AAPD, 2020. (4)

Inclusion Criteria:

1. 4 -9 years old
2. Primary molars with no spontaneous or provoked pain
3. Primary molars with at least two-thirds of the root length were still present.
4. Primary molars with no sign of internal or other kinds of root or bone resorption.

Exclusion Criteria:

1. Patients with systemic diseases (congenital or rheumatic heart disease, hepatitis, nephritis, tumor, cyclic neutropenia, leukemia, and children on long-term corticosteroid therapy).
2. Un-cooperative patients.
3. Un-restorable primary molars (Grossly broken-down primary molars that have decay extending way under the gingiva and tooth with root caries).

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success | (at 3,6,9and 12 months)
  • Success clinically and radiographically will assess by the number of participants with symptoms-free and no peri-radicular pathology

CONTACTS AND LOCATIONS:
Locations (1):
- MSA University, El-Sheikh Zayed City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided